CLINICAL TRIAL: NCT00162175
Title: A Phase 3, Randomized, Double-blind, Placebo Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of BMS-298585 in Combination With Glyburide Therapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Sulfonylurea Therapy Alone
Brief Title: PPAR-COMBO With Sulfonylurea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV168-021
Record Dates: First submitted 2005-09-09; First posted 2005-09-13 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2007-09

CONDITIONS: Metabolics Diabetes Nos
MeSH Terms: interventions — muraglitazar

INTERVENTIONS:
Drug: Muraglitazar

SUMMARY:
A Phase 3, Randomized, Double-blind, Placebo Controlled, Multicenter Trial to Evaluate the Safety and Efficacy of BMS-298585 in Combination with Glyburide Therapy in Subjects with Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Sulfonylurea Therapy Alone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes, HbA1c > 7.0% and < 10.0%, mean serum triglyceride < 600 mg/dL, body mass index < 41 kg/m2, fasting c-peptide . 1.5 ng/mL.

Exclusion Criteria:

* History of MI (myocardial infarction), coronary angioplasty or bypass graft(s), valvular disease or repair, unstable angina pectoris, transient ischemic attack (TIA), cerebrovascular attack, or cerebrovascular accident (CVA) within 6 months, congestive heart failure (NYHA Class III and IV, uncontrolled hypertension, history or renal disease, peripheral vascular disease (PVD), pulmonary disease, gastrointestinal disease, active liver disease or endocrine disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534
Dates: Start 2003-07; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Compare change from baseline in HbA1c after 24 weeks of treatment with muraglitazar + glyburide vs placebo + glyburide

SECONDARY OUTCOMES:
Change in FPG from basline to W24, proportion of subjects receiving therapeutic response at W24, percent change of fasting lipid levels from baseline to W11/12, change in hs-CRP from baseline to W24

CONTACTS AND LOCATIONS:
Locations (149):
- United States (74):
  - Local Institution, Anniston, Alabama
  - Local Institution, Hoover, Alabama
  - Local Institution, Huntsville, Alabama
  - Local Institution, Mobile, Alabama
  - Local Institution, Mesa, Arizona
  - Local Institution, Phoenix, Arizona
  - Local Institution, Tucson, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Encinitas, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Mission Viejo, California
  - Local Institution, Pasadena, California
  - Local Institution, San Diego, California
  - Local Institution, Walnut Creek, California
  - Local Institution, Westlake Village, California
  - Local Institution, Colorado Springs, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Loveland, Colorado
  - Local Institution, Wheat Ridge, Colorado
  - Local Institution, Chipley, Florida
  - Local Institution, Miami, Florida
  - Local Institution, New Port Richey, Florida
  - Local Institution, Pinellas Park, Florida
  - Local Institution, Vero Beach, Florida
  - Local Institution, Winter Park, Florida
  - Local Institution, Dunwoody, Georgia
  - Local Institution, Chicago, Illinois
  - Local Institution, Overland Park, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Slidell, Louisiana
  - Local Institution, Chester, Maryland
  - Local Institution, Silver Springs, Maryland
  - Local Institution, Springfield, Massachusetts
  - Local Institution, Berkley, Michigan
  - Local Institution, Detroit, Michigan
  - Local Institution, Arden Hills, Minnesota
  - Local Institution, Gulfport, Mississippi
  - Local Institution, Excelsior Springs, Missouri
  - Local Institution, Kansas City, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, East Syracuse, New York
  - Local Institution, Charlotte, North Carolina
  - Local Institution, Greensboro, North Carolina
  - Local Institution, Hickory, North Carolina
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Morehead City, North Carolina
  - Local Institution, Wilmington, North Carolina
  - Local Institution, Cincinnati, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Corvallis, Oregon
  - Local Institution, Eugene, Oregon
  - Local Institution, Portland, Oregon
  - Local Institution, Altoona, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Cranston, Rhode Island
  - Local Institution, Anderson, South Carolina
  - Local Institution, Duncan, South Carolina
  - Local Institution, Simpsonville, South Carolina
  - Local Institution, Summerville, South Carolina
  - Local Institution, Bristol, Tennessee
  - Local Institution, Kingsport, Tennessee
  - Local Institution, Knoxville, Tennessee
  - Local Institution, Memphis, Tennessee
  - Local Institution, Dallas, Texas
  - Local Institution, Houston, Texas
  - Local Institution, Irving, Texas
  - Local Institution, Lake Jackson, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, The Colony, Texas
  - Local Institution, Olympia, Washington
  - Local Institution, Bluefield, West Virginia
  - Local Institution, Marshfield, Wisconsin
- Argentina (5):
  - Local Institution, Bahía Blanca, Buenas Aires
  - Local Institution, Buenos Aires, Buenos Aires
  - Local Institution, Capital Federal, Buenos Aires
  - Local Institution, Córdoba, Córdoba Province
  - Local Institution, Mendoza, Mendoza Province
- Australia (3):
  - Local Institution, Canberra, New South Wales
  - Local Institution, Wollongong, New South Wales
  - Local Institution, Brisbane, Queensland
- Brazil (4):
  - Local Institution, Curitiba, Paraná
  - Local Institution, Belém, Pará
  - Local Institution, Porto Alegre, Rio Grande do Sul
  - Local Institution, Marília, São Paulo
- Canada (7):
  - Local Institution, Corunna, Ontario
  - Local Institution, Hawksbury, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Gatineau, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Saint-Jérôme, Quebec
  - Local Institution, St. John's
- France (6):
  - Local Institution, Rosiers, D'Egletons
  - Local Institution, Labarthe, Sur Leze
  - Local Institution, Husseren-Wesserling, Wesserling
  - Local Institution, Broglie
  - Local Institution, Chartres
  - Local Institution, Gémenos
- Germany (4):
  - Local Institution, Viernheim, Schwenningen
  - Local Institution, Dresden
  - Local Institution, Hamburg
  - Local Institution, Nuremberg
- Local Institution, Ravenna, Italy
- Mexico (7):
  - Local Institution, Durango, Durango
  - Local Institution, Tijuana, Estado de Baja California
  - Local Institution, León, Guanajuato
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Alburquerque, New Mexico
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Mérida, Yucatán
- Netherlands (6):
  - Local Institution, Deurne
  - Local Institution, Ewyk
  - Local Institution, Hoogvliet
  - Local Institution, Rijswijk
  - Local Institution, The Hague
  - Local Institution, Zwijndrecht
- Peru (2):
  - Local Institution, Arequipa, Arequipa
  - Local Institution, Lima, Lima Province
- Puerto Rico (4):
  - Local Institution, Carolina
  - Local Institution, Guaynabo
  - Local Institution, Ponce
  - Local Institution, Rio Piedras
- Russia (4):
  - Local Institution, Moscow
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Smolensk
- Spain (11):
  - Local Institution, Santiago, De Compostela
  - Local Institution, Las Palmas, DE
  - Local Institution, A Coruña
  - Local Institution, Alicante
  - Local Institution, Cadiz
  - Local Institution, Granada
  - Local Institution, Madrid
  - Local Institution, Oviedo
  - Local Institution, Santa Cruz de Tenerife
  - Local Institution, Teruel
  - Local Institution, Zaragoza
- United Kingdom (11):
  - Local Institution, Soham, Cambridgeshire
  - Local Institution, Bexhill-on-Sea, East Sussex
  - Local Institution, Sunbury-on-Thames, Greater London
  - Local Institution, Aldershot, Hampshire
  - Local Institution, Glasgow, Lanarkshire
  - Local Institution, Blackpool, Lancashire
  - Local Institution, Harrow, Middlesex
  - Local Institution, Hastings, Sussex
  - Local Institution, Bath, Wiltshire
  - Local Institution, Inkberrow, Worcestershire
  - Local Institution, Swan Lane

REFERENCES:
- [Derived] Rubin CJ, De Pril V, Fiedorek FT. Coadministration of muraglitazar plus glyburide: improvement of glycaemic and lipid profiles in patients with type 2 diabetes. Diab Vasc Dis Res. 2009 Apr;6(2):120-32. doi: 10.1177/1479164109336049. PMID 20368202